CLINICAL TRIAL: NCT01834027
Title: The Effect of Jazz on Postoperative Pain and Stress in Patients Undergoing Elective Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Sonia Vaida, Professor of Anesthesiology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 40925
Record Dates: First submitted 2012-11-30; First posted 2013-04-17 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-03

CONDITIONS: Pain; Anxiety
Keywords: music; stress; anxiety; post-surgical; pain
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Jazz music (Experimental): Jazz music will be played through headphones to post-surgical hysterectomy patients while they are in the post anesthesia care unit.
  Interventions: Behavioral: Jazz music
- No music (Active Comparator): The patients in this group with have headphones but no music will be played.
  Interventions: Behavioral: No music

INTERVENTIONS:
Behavioral: Jazz music — Jazz music from artists including Miles Davis, Ella Fitzgerald, Nat King Cole, Dave Brubeck, etc. will be played through headphones for post-surgical hysterectomy patients while they are in the post anesthesia care unit.
  Arms: Jazz music
Behavioral: No music — In this group no music will be played in PACU
  Other Names: control group
  Arms: No music

SUMMARY:
The purpose of this study is to investigate the effects of music on patients after surgery in the Post Anesthesia Care Unit (PACU). For many patients, surgery creates significant emotional stress and anxiety which can include discomfort or pain. Music therapy has proven to be a useful adjuvant in various inpatient and outpatient settings by providing a relaxing effect that decreases heart rate, blood pressure, and hormonal measures of stress. It has been shown that classical music can cause physiological and psychological differences in patient outcomes, but few studies have looked specifically at effects of jazz music. Some have argued that jazz may be too involved to provide the same relaxed state as classical music, but this may be due in part to the type of jazz played for the patient. It is our hypothesis that slow jazz music by artists including Miles Davis, Ella Fitzgerald, Diana Krall, Dave Brubeck, etc. will reduce measures of stress and anxiety in patients in the PACU following surgery for hysterectomy (laparoscopic or robotic) to a greater extent than the control group. Jazz music or "no music" will be played through headphones to participants in the study post-surgically while they are in the PACU and measures of stress, anxiety, and pain will be monitored.

DETAILED DESCRIPTION:
* Patients will be identified the morning of surgery from the operating room schedule.
* The patients will be randomized to two groups: jazz music or no music.
* Head phones will be applied to all patients included in the study; in one group jazz music will be provided through the headphones. The second group no music will be played.
* Blood pressure will be monitored by a non-invasive blood pressure cuff at 5 minute intervals throughout the patient's stay in the PACU.
* Heart rate will be measured, using a pulse oximeter, at the same intervals as blood pressure.
* Before the patient leaves the PACU, she will be asked to rate her perception of her levels of pain and anxiety on scales that use a numeric scale of 1-10. The primary variable outcomes are: heart rate and mean blood pressure. Secondary outcomes include: perceived pain, anxiety, and level of relaxation.
* headphones will be used to deliver one of the following sounds to the patients: 1) jazz music (BPM<100) by artists including Miles Davis, Ella Fitzgerald, Diana Krall, Dave Brubeck, etc.; or 2) no music providing.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective hysterectomy (laparoscopic or robotic)
* ASA 1 or 2
* Normotensive
* Normal heart rate

Exclusion Criteria:

* Patient does not wish to participate in the study
* Deaf or hearing impaired patients
* Ear deformities or abnormalities
* Pre-existing diagnosis of anxiety disorder, depression, substance abuse, or any other psychiatric diagnoses

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Vaida, MD, Principal Investigator — Penn State University; Jansie Prozesky, MD, Principal Investigator — Penn State University
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- No Music: The patients in this group with have headphones but no music will be played.
  No music: In this group nu music will be played in PACU
Period: Overall Study
Arm/Group | Jazz Music | No Music
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The statistical plan and sample size justification were based on the results of a previous study (Nilsson, U. Heart Lung 2009;38(3):201-207) comparing the change in heart rate from pre- to post-surgery between a music and control group.
Groups:
- Jazz Music: Jazz music will be played through noise-cancelling headphones to post-surgical hysterectomy patients while they are in the post anesthesia care unit.
  Jazz music: Jazz music from artists including Miles Davis, Ella Fitzgerald, Nat King Cole, Dave Brubeck, etc. will be played through headphones for post-surgical hysterectomy patients while they are in the post anesthesia care unit.
- No Music: The patients in this group will have noise-cancelling headphones but no music will be played.
  No music: In this group, noise-cancelling headphones will be worn, but no music will be played in PACU
- Total: Total of all reporting groups
Arm/Group | Jazz Music | No Music | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Customized [Number; unit: participants]
  <18 years of age | 0 | 0 | 0
  >=18 and <=75 years | 28 | 28 | 56
  > 75 years of age | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change in Heart Rate From Baseline on Arrival in PACU
Description: Mean difference in heart rate from baseline measurement taken upon the patient's arrival to the PACU. Heart rate will be measured through pulse oximetry
Time Frame: 5, 10, 15, 20, 25, 30 minutes after baseline measurement on patient's arrival in PACU
Measure: Mean (95% Confidence Interval); unit: beats per minute
Arm/Group | Jazz Music | No Music
Number analyzed (Participants) | 28 | 28
beats per minute
  5 minutes after baseline measurement | -3.39 [-7.03 to -0.25] | -5.11 [-8.75 to -1.47]
  10 minutes after baseline measurement | -4.18 [-8.37 to 0.02] | -4.71 [-8.91 to -0.52]
  15 minutes after baseline measurement | -5.21 [-9.67 to -0.75] | -6.46 [-10.93 to -1.98]
  2- minutes after baseline measurement | -6.29 [-11.23 to -1.34] | -6.61 [-11.57 to -1.66]
  25 minutes aqfter baseline measurement | -6.68 [-11.57 to -1.79] | -8.58 [-13.49 to -3.67]
  30 minutes after baseline measurement | -5.71 [-10.74 to -0.96] | -5.36 [-10.11 to -0.60]

2. Secondary Outcome: Difference in Patient's Perception of Anxiety From Baseline Score Upon Arrival in the PACU
Description: Upon arrival in the PACU, patient will be asked to rate her level of anxiety using a numeric rating scale from 0-10 (0 indicates no anxiety while 10 indicates extreme anxiety). After wearing headphones for 30 minutes, with either jazz music or no music, the patient will reassess her anxiety level. The difference between the 30 minute score and the baseline will be calculated.
Time Frame: Once, at 30 minutes after the patient entered the PACU
Population: 2 participants in the jazz group nad 1 participant in the no music group did not provide an anxiety score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Jazz Music | No Music
Number analyzed (Participants) | 26 | 27
units on a scale | 0.1 (0.92) | 0 (0.43)

3. Secondary Outcome: Mean Difference in Patient's Perception of Pain From Baseline
Description: The patient will be asked to rate her level of pain using a numeric rating scale from 0-10 (0 indicates no pain and 10 indicates extreme pain). Baseline will be value upon entering PACU. The difference between the values at specific times and the baseline value will be calculated.
Time Frame: 10, 20 , and 30 minutes after baseline measurement
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Jazz Music | No Music
Number analyzed (Participants) | 28 | 28
units on a scale
  10 minutes after baseline measurement | 1.04 [-0.28 to 2.35] | -0.95 [-2.31 to 0.40]
  20 minutes after baseline measurement | 0.61 [-0.80 to 2.02] | -0.16 [-1.61 to 1.28]
  30 minutes after baseline measurement | 0.77 [-0.83 to 2.36] | -.03 [-1.92 to 1.33]

4. Secondary Outcome: Mean Blood Pressure
Description: non-invasive mean blood pressure will be measured every 5 minutes for a period of 60 minutes
Time Frame: 60 minutes
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Jazz Music | No Music
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No